CLINICAL TRIAL: NCT04158843
Title: A Randomized, Open Label Trial to Evaluate Radical Local Treatment Versus Palliative Treatment for Breast Cancer Patients With Ipsilateral Humerus or Sternum Oligometastasis
Brief Title: Radical Local vs. Palliative Therapy for Breast Cancer Patientts With Ipsilateral Humerus or Sternum Oligometastasis
Acronym: BOMB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: xuexin he (Other)
Responsible Party: Sponsor-Investigator, xuexin he, Associate chief physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOMB
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer; Oligometastasis
Keywords: Breast Cancer; Oligometastasis; Humerus; Sternum
MeSH Terms: conditions — Breast Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radical local treatment (Experimental): Radical resection is performed, and the cutting edge is negative, or radical local radiotherapy is feasible (cumulative radiotherapy dose is greater than or equal to 50Gy). Systemic endocrine therapy and targeted therapy are allowed after radical local therapy. However, whether systemic chemotherapy should be used is determined by clinicians according to clinical experience or guidelines.
  Interventions: Procedure: Radical resection; Radiation: Radical radiotherapy
- Palliative treatment (Active Comparator): No radical surgical resection or radical surgical resection or radiotherapy is performed in this group. But palliative internal fixation or radiotherapy for pain relief is permitted. Moreover, systemic chemotherapy, endocrine therapy and targeted therapy are allowed.
  Interventions: Other: Palliative treatment

INTERVENTIONS:
Procedure: Radical resection — Radical resection is performed, and the cutting edge is negative.
  Arms: Radical local treatment
Radiation: Radical radiotherapy — Radical local radiotherapy is feasible (cumulative radiotherapy dose is greater than or equal to 50Gy).
  Arms: Radical local treatment
Other: Palliative treatment — Including palliative internal fixation, radiotherapy, systemic chemotherapy, endocrine therapy or targeted therapy
  Arms: Palliative treatment

SUMMARY:
A Randomized, Open Label, Phase III Trial to Evaluate Radical Local Treatment versus Palliative Treatment for Breast Cancer Patients with Primary Ipsilateral Humerus or Sternum Oligometastasis

DETAILED DESCRIPTION:
This is a prospective, randomized, and multicenter study to compare the radical local treatment versus palliative treatment for breast cancer patients with primary ipsilateral humerus or sternum oligometastasis.

183 subjects will be randomized divided into two groups (experimental group and control group) at a ratio of 2 to 1.

Control group: Palliative treatment. No radical surgical resection or radiotherapy is performed in this group. But palliative internal fixation or radiotherapy for pain relief is permitted. Moreover, systemic chemotherapy, endocrine therapy and targeted therapy are allowed.

Experimental group：Radical local treatment. Radical resection is performed, and the cutting edge is negative, or radical local radiotherapy is feasible (cumulative radiotherapy dose is greater than or equal to 50Gy). Systemic endocrine therapy and targeted therapy are allowed after radical local therapy. However, whether systemic chemotherapy should be used is determined by clinicians according to clinical experience or guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients provided written informed consent
* Women aged 18-75 years old
* Histologically confirmed breast cancer and after radical mastectomy
* Patients of breast cancer with ipsilateral humerus or sternum oligometastasis, and there is no imaging evidence of other site metastases
* Patients must have recovered to baseline condition or to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade = 1 from any acute CTCAE v. 5.0 grade =2 side effects of previous treatments
* Without infection of human immunodeficiency virus (HIV) on central laboratory assay results prior to randomization
* Alanine aminotransferase (ALT) </= 2.5 × the upper limit of normal (ULN), Aspartate aminotransferase (AST) </= 2.5 × ULN prior to randomization
* Total bilirubin (TBIL) </= 1.25 × ULN
* Alkaline phosphatase (ALK) </= 2.5 × ULN
* Gamma glutamyl transpeptidase (GGT) </= 2.5 × ULN
* Albumin >/= 30g/L
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2
* Women of child-bearing age should take effective contraceptive measures
* Serum total bilirubin (TBil) </= 1.5 × ULN
* Serum creatinine (Scr) </= 1.5 × ULN
* White blood cell count (WBC) >/= 3×109/L, Blood neutrophil count >/= 1.5×109/L, Platelet count >/= 100×109/L, Hemoglobin (HB) >/= 9 g/dL

Exclusion Criteria:

* Without radical mastectomy of the primary breast lesions
* No radical resection or radiotherapy is possible for metastatic lesions
* Other site metastases except ipsilateral humerus or sternum are present
* With multiple metastatic lesions
* Any other current malignancy or malignancy diagnosed within the past five years (other than carcinoma in situ or stage Ia carcinoma of the cervix, skin basal cell carcinoma and papillary thyroid carcinoma at early stage)
* Active infection with human immunodeficiency virus (HIV) prior to first study treatment administration.
* History of participating any other clinical trials within 30 days prior to randomization
* Known unable to tolerate humerus or sternal surgery or radical radiotherapy
* Pregnancy or lactation
* Current severe systemic disease (for example, clinically significant cardiovascular, pulmonary, or renal disease)
* Legal incompetence or limitation.
* Considered unable to complete the study or sign the informed consent due to a medical or mental disorder by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2020-05-09 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 4 years
  PFS is defined as time from randomization to disease progression or death, whichever occurs first

SECONDARY OUTCOMES:
Overall Survival (OS) | 4 years
  OS is defined as time from randomization to death for any cause. If there is no death reported for a subject before the date cutoff for OS analysis, OS will be censored at the last contact date at which the subject is known to be alive.
  For patients who had not died up to the cut-off date, the date they were last known to be alive was derived from the patient status records, the trial completion record, radiological imaging assessments, the study treatment termination record, and the randomization date.
Patient Reported Outcomes | 4 years
  Breast cancer specific health treatment related quality of life and general health status (Functional Assessment of Cancer Therapy-Breast (FACT-B) [version 4])

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobo Yan, MD, Study Director — The Second Affiliated Hospital of Zhejiang University School of Medicidne
Locations (4):
- China (4):
  - Institute of Cancer Research and Basic Medical Sciences, CAS Cancer Hospital, University of Chinese Academy of Sciences Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine (SAHZU), Hangzhou, Zhejiang
  - Jiaxing Second Hospital, Jiaxing, Zhejiang
  - The Central Hospital of Lishui, Lishui, Zhejiang